CLINICAL TRIAL: NCT00555152
Title: Neoadjuvant Trial of Lapatinib for the Treatment of Women With DCIS Breast Cancer
Brief Title: Lapatinib Ditosylate in Treating Patients With Ductal Breast Carcinoma In Situ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCI-2009-00875; NCI-2009-00875 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2008-0086; NCT00570453; CDR0000573719; H-19895; P50CA058183 (NIH); P30CA016672 (NIH); NCT00570453 (obsolete NCT alias)
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-03

CONDITIONS: Ductal Breast Carcinoma In Situ; HER2/Neu Positive
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Lapatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (lapatinib ditosylate) (Experimental): Patients receive lapatinib ditosylate PO once QD for 2-6 weeks until the time of surgery.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lapatinib Ditosylate
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD for 2-6 weeks until the time of surgery.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lapatinib Ditosylate — Given PO
  Other Names: Tykerb
  Arms: Arm I (lapatinib ditosylate)
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)

SUMMARY:
This randomized phase I/II trial studies the side effects and best dose of lapatinib ditosylate and to see how well it works in treating patients with ductal breast carcinoma in situ. Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether lapatinib (lapatinib ditosylate) therapy at the dose of 1000 mg results in a statistically significantly lower rate of proliferation in ductal carcinoma in situ (DCIS) breast cancer cells as measured by Ki67 when compared to placebo.

II. Determine the toxicity profile and frequency of adverse events in women with DCIS breast cancer taking lapatinib at 1000 mg as compared to women taking placebo.

SECONDARY OBJECTIVES:

I. Determine whether lapatinib treatment affects the incidence of DCIS seen at the time of surgical excision.

II. Determine whether treatment with lapatinib will modulate breast tissue histology or the expression of specific biomarkers in normal and DCIS breast cancer cells.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive lapatinib ditosylate orally (PO) once daily (QD) for 2-6 weeks until the time of surgery.

ARM II: Patients receive placebo PO QD for 2-6 weeks until the time of surgery.

After completion of study treatment, patients are followed for 4-5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be premenopausal or postmenopausal
* Participants must have a diagnosis of ductal carcinoma in situ made by core needle biopsy
* The DCIS cells must have high expression of human epidermal growth factor receptor 2 (erbB2) (3+ by immunohistochemical staining or amplification by fluorescence in situ hybridization [FISH]), and/or have detectable expression of epidermal growth factor receptor (EGFR) (1+ or more by immunohistochemical staining)
* All participants must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* Individuals with a diagnosis of breast cancer, non-melanoma skin cancer, cervical cancer in situ, or early bladder cancer are eligible if they have not been treated with chemotherapy, biological therapy, or breast radiotherapy to the breast currently affected by DCIS within one year; in addition, individuals with a diagnosis of breast cancer may not have used tamoxifen, raloxifene, or other antiestrogen compounds within three months of study day 1
* If subjects are of reproductive potential, they must agree to use a reliable contraceptive method or be sexually abstinent; subjects must fulfill these conditions beginning at the time of starting study medications and ending one month after study termination
* Negative serum pregnancy test (beta-human chorionic gonadotropin [HCG]) at baseline (within 30 days of day 0) for women of child bearing potential
* Serum creatinine =< 1.5 times the institution?s upper limit of normal
* Total bilirubin =< 1.5 times the institution's upper limits of normal
* Serum glutamic oxaloacetic transaminase (SGOT) =< 1.5 times the institution's upper limits of normal
* Alkaline phosphatase =< 1.5 times the institution's upper limits of normal
* Albumin =< 1.5 times the institution's upper limits of normal
* White blood cells (WBC) > 4.0 k/uL
* Platelet count > 100,000/uL
* Hematocrit of > 30%
* Cardiac ejection fraction within normal limits for the institution by multi gated acquisition scan (MUGA) scan or normal cardiac ultrasound (defined as within the upper limit of normal [ULN] for the institution)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Willingness to refrain from donating blood to others during the study

Exclusion Criteria:

* Individuals are ineligible if they have either active cancer or a prior history of malignancies other than (e.g., breast cancer, skin cancer [basal or squamous cell carcinoma], cervical cancer in situ, or early bladder cancer [preinvasive transitional cell carcinoma of the bladder]) within the past five years
* Participants are ineligible if they are currently being treated with tamoxifen, raloxifene, or with aromatase inhibitors (letrozole, anastrozole, exemestane)
* Individuals are ineligible if they have received chemotherapy, biological therapy (e.g., Herceptin), or radiotherapy for the treatment of any cancer within 1 year or if they have received tamoxifen, raloxifene, letrozole, anastrozole, or exemestane therapy within 3 months of study day 1
* Individuals currently receiving anticoagulation therapy (e.g., Coumadin) are ineligible
* Blood urea nitrogen [BUN] > 1.5 x ULN or
* Creatinine [Cr] > 1.5 x ULN
* SGOT > 1.5 x ULN
* Serum glutamate pyruvate transaminase (SGPT) > 1.5 x ULN
* Alkaline phosphatase > 1.5 x ULN
* Bilirubin > 1.5x ULN
* Individuals who are currently participating in a study of an investigational drug
* Pregnancy, lactation or unwillingness to use a reliable contraceptive method in women of childbearing potential
* Severe underlying chronic illness or disease, such as uncontrolled diabetes
* Individuals with known congestive heart disease or previous myocardial infarction are ineligible
* Patients taking any prohibited medications
* Individuals with hypokalemia or hypomagnesemia are ineligible unless these conditions are corrected to within normal limits before starting drug
* Individuals with congenital long QT syndrome or baseline QTcF intervals > 480 msec on electrocardiogram (EKG)
* Individuals taking anti-arrhythmics, beta blockers, or other medications that may lead to QT prolongation
* Individuals who have received a cumulative dose of anthracycline therapy greater than 500 mg/m^2 are ineligible

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-08-19 (Actual); Primary Completion 2014-08-28 (Actual); Study Completion 2014-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Powel Brown, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Activated 1/17/2008 at Baylor College of Medicine (BCM), MD Anderson Cancer Center, Dana-Farber Cancer Institute, Mayo Clinic, Georgetown University & Walter Reed Army Medical Center; closed at BCM 3/8/2010, re-activated 9/19/2011 at MD Anderson, Dana-Farber Cancer Institute, Mayo Clinic & University of Alabama, Birmingham, closed 8/28/2014.
Pre-assignment Details: A total of 22 participants were enrolled and randomized to 3 of 4 treatment arms; Two of the 4 initial arms were removed in the second period with one of those having no enrollment. Three participants were enrolled while the study was open at BCM, the other 19 were enrolled after the study was transferred to MD Anderson (second study period).
Groups:
- Arm I Lapatinib 1500 mg: Lapatinib ditosylate 1500 mg orally once daily for 2-6 weeks until the time of surgery.
- Arm II Lapatinib 1000 mg: Lapatinib 1000 mg orally once daily for 2-6 weeks until the time of surgery.
- Arm III Lapatinib 750 mg: Lapatinib 750 mg orally once daily for 2-6 weeks until the time of surgery.
- Arm IV Placebo: Placebo orally once daily for 2-6 weeks until the time of surgery.
Period: Period Open at BCM: 1/17/08-3/8/10
Arm/Group | Arm I Lapatinib 1500 mg | Arm II Lapatinib 1000 mg | Arm III Lapatinib 750 mg | Arm IV Placebo
Started | 2 | 0 (Participants in initial and second study registration periods reported separately.) | 0 | 1
Completed | 2 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0
Period: Transfer to MD Anderson: 9/19/11-8/28/14
Arm/Group | Arm I Lapatinib 1500 mg | Arm II Lapatinib 1000 mg | Arm III Lapatinib 750 mg | Arm IV Placebo
Started | 0 (Participants in initial and second study registration periods reported separately.) | 10 | 0 | 9
Completed | 0 | 10 | 0 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I Lapatinib 1500 mg | Arm II Lapatinib 1000 mg | Arm III Lapatinib 750 mg | Arm IV Placebo | Total
Number analyzed (Participants) | 2 | 10 | 0 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (9.5) | 51.7 (10.7) |  | 52 (8.4) | 51.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 10 |  | 10 | 22
  Male | 0 | 0 |  | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 |  | 2 | 3
  Not Hispanic or Latino | 2 | 9 |  | 8 | 19
  Unknown or Not Reported | 0 | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0 | 0
  Asian | 0 | 1 |  | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0 | 0
  Black or African American | 0 | 0 |  | 0 | 0
  White | 2 | 9 |  | 9 | 20
  More than one race | 0 | 0 |  | 0 | 0
  Unknown or Not Reported | 0 | 0 |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 10 |  | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Proliferation (Ki67 IHC) in Ductal Breast Carcinoma In Situ (DCIS)
Description: Reduction in percent of Ki67 positive cells at surgery compared to baseline as a function of treatment. Analysis of the primary treatment comparison will be based on a two sample t-test comparing change in log-transformed Ki67% for placebo and treated subjects. P-values of 0.05 will be considered significant. Proliferation will be assessed by immunohistochemical (IHC) staining for Ki67, and the change in percentage of Ki67 positive cells will be compared in lapatinib-treated samples versus placebo.
Time Frame: 2-6 weeks from baseline to surgery, up to 6 weeks
Population: No outcome data available due to laboratory issues affecting the analysis of biomarkers results.
Arm/Group | Arm I Lapatinib 1500 mg | Arm II Lapatinib 1000 mg | Arm III Lapatinib 750 mg | Arm IV Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Incidence of Ductal Carcinoma in Situ Remaining at Resection
Description: Number of participants with DCIS incidence on surgical excision. Differences in histologic response (disappearance of DCIS) will be evaluated using Fisher's exact test. Correlation analysis and linear models will be used to evaluate associations among marker values at baseline and among changes in marker values and treatment. All statistical tests will be two-sided.
Time Frame: 2-6 weeks from baseline to surgery, up to 6 weeks
Population: DCIS was present at the time of surgery in all patients.
Measure: Number; unit: participants
Arm/Group | Arm I Lapatinib 1500 mg | Arm II Lapatinib 1000 mg | Arm III Lapatinib 750 mg | Arm IV Placebo
Number analyzed (Participants) | 2 | 10 | 0 | 10
participants
  Present | 2 | 10 |  | 10
  Absent | 0 | 0 |  | 0
Statistical Analysis 1: Comparison: Arm I Lapatinib 1500 mg vs Arm II Lapatinib 1000 mg vs Arm III Lapatinib 750 mg vs Arm IV Placebo; Test type: Superiority or Other; p = 1, Fisher Exact

3. Secondary Outcome: Biomarker Analysis of Proliferation Markers
Description: Correlation analysis and linear models will be used to evaluate associations among marker values at baseline and among changes in marker values and treatment. All statistical tests will be two-sided.
Time Frame: 2-6 weeks from baseline to surgery, Up to 6 weeks
Population: No outcome data available due to laboratory issues affecting the analysis of biomarkers results.
Arm/Group | Arm I Lapatinib 1500 mg | Arm II Lapatinib 1000 mg | Arm III Lapatinib 750 mg | Arm IV Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Primary Outcome: Incidence of Adverse Events Graded According to the National Cancer Institute (NCI) Common Terminology Criteria (CTCAE) Version 3.0
Description: Toxicity profile summarized reflects incidence by number of participants affected with adverse events by Maximum Grade 1 to 3, additional adverse event according to the NCI CTCAE version 3.0 reported in Adverse Event section results.
Time Frame: From baseline to 4-5 weeks after surgery
Measure: Number; unit: participants
Arm/Group | Arm I Lapatinib 1500 mg | Arm II Lapatinib 1000 mg | Arm III Lapatinib 750 mg | Arm IV Placebo
Number analyzed (Participants) | 2 | 10 | 0 | 10
participants
  Grade 3 | 0 | 0 |  | 1
  Grade 2 | 2 | 6 |  | 3
  Grade 1 | 0 | 3 |  | 4

ADVERSE EVENTS:
Time Frame: Subjects followed up to 4-5 weeks after surgery to assess for adverse events with overall collection period approximately five years, first study period January 2008 to March 2010 and second September 2011 to August 2014.
Arm/Group | Arm I Lapatinib 1500 mg | Arm II Lapatinib 1000 mg | Arm III Lapatinib 750 mg | Arm IV Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/10 | 0/0 | 1/10
Other Adverse Events (participants affected / at risk) | 2/2 | 9/10 | 0/0 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I Lapatinib 1500 mg (N=2) | Arm II Lapatinib 1000 mg (N=10) | Arm III Lapatinib 750 mg (N=0) | Arm IV Placebo (N=10)
Hematoma (Vascular disorders) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1 — Infection with normal absolute neutrophil count (ANC) or grade 1 or 2 neutrophils
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I Lapatinib 1500 mg (N=2) | Arm II Lapatinib 1000 mg (N=10) | Arm III Lapatinib 750 mg (N=0) | Arm IV Placebo (N=10)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 | 2 | 0 | 0
Constitutional Symptoms (General disorders) | 0 | 1 | 0 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 | 2 | 0 | 1
Insomnia (General disorders) | 1 | 0 | 0 | 0
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0
Flushing (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 2
Hot flashes/flushes (Endocrine disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Dehydration (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 7 | 0 | 2
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Mucositis/stomatitis (clinical exam) Oral cavity (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 4 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Hemorrhage, GI Rectum (Vascular disorders) | 0 | 1 | 0 | 0
Hemorrhage, GU Vagina (Vascular disorders) | 1 | 0 | 0 | 0
Hemorrhage, pulmonary/upper respiratory Nose (Vascular disorders) | 1 | 0 | 0 | 0
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Vascular disorders) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Lymphatics (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 1
Neuropathy: sensory (Nervous system disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 3 | 0 | 2
Pain -Other (General disorders) | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary/Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Bladder spasms (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal/Genitourinary (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cytokine release syndrome/acute infusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less